CLINICAL TRIAL: NCT03794089
Title: Reducing Anxiety and Stress in Primary Care Patients: Pilot RCT of a Brief Intervention (CDA 15-262)
Brief Title: Reducing Anxiety and Stress in Primary Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CDX 18-006
Record Dates: First submitted 2019-01-02; First posted 2019-01-04 (Actual); Results first posted 2022-06-07 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Anxiety
Keywords: anxiety; primary health care; Veterans
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial with randomization to the intervention condition or control condition
Who Masked: Outcomes Assessor
Masking Description: Baseline assessment, monthly follow-up assessments, and post assessment will be conducted by research assistants who are masked to participant condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brief anxiety intervention (Experimental): Modular anxiety intervention designed for PC-MHI, up to six 30-minute sessions occurring approximately every 2 weeks, patients select modules of interest to them to complete, emphasis on psycho-education and cognitive-behavioral coping strategies for self-management
  Interventions: Behavioral: Brief anxiety intervention
- Usual PC-MHI care (Active Comparator): Appointment with PC-MHI provider at local primary care clinic, providers delivers whatever interventions they deem appropriate and collaboratively decides with patients whether and when to meet again as in routine PC-MHI care
  Interventions: Behavioral: Usual PC-MHI care

INTERVENTIONS:
Behavioral: Brief anxiety intervention — Modular anxiety intervention, tailored for Veterans, with emphasis on adaptive coping skills
  Arms: Brief anxiety intervention
Behavioral: Usual PC-MHI care — Anxiety treatment with mental health provider in local primary care clinic
  Arms: Usual PC-MHI care

SUMMARY:
Anxiety is common among primary care patients, but is undertreated. The purpose of this study is to evaluate whether a brief anxiety treatment designed for VA primary care is more effective at reducing anxiety symptoms in Veterans compared to usual care. The investigators will also examine whether Veterans like the brief treatment and whether the treatment can be feasibly delivered in primary care. Forty-eight adult Veteran primary care patients from the Syracuse VAMC who are experiencing anxiety symptoms will be recruited and randomly assigned to receive the brief anxiety treatment or usual care. The brief treatment consists of up to six 30-minute sessions with a cognitive-behavioral skills focus. The investigators will compare anxiety symptom severity between the two groups at baseline and at post-assessment 16 weeks later.

DETAILED DESCRIPTION:
Background/Rationale: Many Veteran primary care patients experience impairing symptoms of anxiety, but rates of treatment are low. Primary Care-Mental Health Integration (PC-MHI), in which mental health clinicians provide brief treatment in the primary care setting, can bridge the gap between demand for, and availability of, anxiety treatment. However, brief anxiety interventions suitable for use in the PC-MHI setting are needed. Developing an effective brief PC-MHI intervention for anxiety would address a gap in VA treatment options and facilitate high quality healthcare that improves treatment engagement, clinical outcomes, and patient experience. To ensure maximum reach, this intervention should accommodate a variety of subthreshold and diagnostic anxiety presentations, as well as comorbid depression.

Objectives: The overall goal of this research program is to develop, refine, and evaluate a brief anxiety intervention that will be acceptable to Veterans and feasible for PC-MHI providers. The primary aim of the current study is to conduct a pilot randomized controlled trial to evaluate feasibility, acceptability, potential implementation barriers and facilitators, and effectiveness of the intervention compared to usual care.

Methods: This will be a pilot hybrid type I effectiveness-implementation randomized controlled trial (N = 35). The primary goal is to evaluate feasibility, acceptability, and effectiveness of the intervention in reducing anxiety symptom severity compared to usual care. The secondary goal is to collect preliminary data on implementation barriers and facilitators that may affect future real-world uptake.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Veteran seen in the Syracuse VA Medical Center primary care clinic in the past year
* Screen positive for current (past 2 weeks) clinically significant anxiety symptoms (8 on Generalized Anxiety Disorder-7)

Exclusion Criteria:

* Inability to communicate in English (as assessed by study staff)
* Report or demonstrate hearing impairment that would preclude telephone screening (as assessed by study staff)
* Inability to demonstrate informed consent

  * defined as not being able to comprehend the study description as assessed by study staff and/or not being able to answer the comprehension of consent questions
  * have a diagnosis of dementia or severe cognitive impairment (defined by primary care provider or self-report, or having a diagnosis in Problem List)
  * screen positive for cognitive impairment (3 or more errors on cognitive screener)
* Have a diagnosis of obsessive-compulsive disorder (OCD) or serious mental illness (SMI) in Problem List

  * i.e., psychotic disorders, bipolar disorder
* Have an encounter diagnosis of post-traumatic stress disorder (PTSD) within the past 2 years OR screen positive for PTSD (3 or more on PC-PTSD-5)
* Currently in psychotherapy/counseling for anxiety and/or depression, defined as any of the following within the past 30 days:

  * attending specialty mental health sessions [excluding a single intake session]
  * attending 2 or more Primary Care-Mental Health Integration sessions
  * Being hospitalized for mental health treatment
* Report severe depressive symptoms (20 or more on Patient Health Questionnaire-9)
* At imminent risk of suicide

  * defined as being identified as imminent risk based on study staff's suicide risk assessment [verified by the PI] and in need of intensive treatment
  * e.g., hospitalization] to ensure safety
* Started or had dosage change in psychotropic medication for anxiety or depression in the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2021-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robyn L. Shepardson, PhD, Principal Investigator — Syracuse VA Medical Center, Syracuse, NY
Locations (1):
- Syracuse VA Medical Center, Syracuse, NY, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shepardson RL, Weisberg RB, Wade M, Maisto SA, Funderburk JS. Brief modular anxiety intervention for primary care: Hybrid I pilot randomized controlled trial of feasibility, acceptability, effectiveness, and implementation potential. J Affect Disord. 2024 Sep 15;361:497-507. doi: 10.1016/j.jad.2024.05.107. Epub 2024 May 27. PMID 38810782

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were adult (age 18 years or older) Veterans recruited from primary care clinics at the Syracuse VA Medical Center from April 2019 through October 2020. Eligible participants were identified through case finding from electronic medical records, direct referrals from primary care and behavioral health providers, or referrals from other local behavioral health research studies.
Pre-assignment Details: A telephone eligibility screening identified those eligible to participate in the study, based on study eligibility criteria including endorsing current anxiety anxiety symptoms and not already being in psychotherapy for anxiety/depression.
Period: Overall Study
Arm/Group | Brief Anxiety Intervention | Usual PC-MHI Care
Started | 17 | 18
Completed 4-week Assessment | 16 | 18
Completed 8-week Assessment | 14 | 18
Completed 12-week Assessment | 13 | 17
Completed | 11 | 17
Not Completed | 6 | 1
Not completed — Lost to Follow-up | 4 | 1
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who completed the Baseline assessment
Groups:
- Total: Total of all reporting groups
Arm/Group | Brief Anxiety Intervention | Usual PC-MHI Care | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.29 (15.76) | 45.56 (16.88) | 47.37 (16.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 15 | 15 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 15 | 16 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 11 | 16 | 27
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 3 | 0 | 3
Generalized Anxiety Disorder-7 [Mean (Standard Deviation); unit: scores on a scale] — Anxiety symptom severity was measured by the Generalized Anxiety Disorder-7 (GAD-7) self-report questionnaire. Participants rate how much they have been bothered by each of 7 anxiety symptoms over the last 2 weeks on a Likert scale from 0 (not at all) to 3 (nearly every day). Scores are summed to create a total score ranging from 0 to 21; higher scores indicate more severe symptoms. The total score is sensitive to change from treatment across the anxiety disorders. The GAD-7 has demonstrated reliability and validity and is a good screening tool for multiple anxiety disorders.
  scores on a scale | 12.76 (4.41) | 11.94 (3.00) | 12.34 (3.72)
Patient Health Questionnaire-9 [Mean (Standard Deviation); unit: scores on a scale] — Depressive symptom severity was measured by the Patient Health Questionnaire-9 (PHQ-9) self-report questionnaire. Participants rate how often they have been bothered by each of 9 symptoms over the last 2 weeks on a Likert scale from 0 (not at all) to 3 (nearly every day). Scores are summed to create a total score from 0 to 27; higher scores indicate greater severity. The total score is sensitive to change from treatment. The PHQ-9 has demonstrated reliability and validity.
  scores on a scale | 11.18 (4.54) | 10.78 (5.08) | 10.97 (4.76)

OUTCOME MEASURES:

1. Primary Outcome: Generalized Anxiety Disorder-7 at Post-Assessment
Description: The primary outcome of anxiety symptom severity will be measured by the Generalized Anxiety Disorder-7 (GAD-7) self-report questionnaire, a validated measure that is widely used in VA primary care. Participants rate how much they have been bothered by each of 7 anxiety symptoms over the last 2 weeks on a Likert scale from 0 (not at all) to 3 (nearly every day). Scores are summed to create a total score ranging from 0 to 21 indicating severity of anxiety symptoms; higher scores indicate more severe symptoms. The total score is sensitive to change from treatment across the anxiety disorders. The GAD-7 has demonstrated reliability and validity and is a good screening tool for multiple anxiety disorders.
Time Frame: Baseline & Post-Assessment (at 16 weeks)
Population: Enrolled participants who completed Post-Assessment at 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Anxiety Intervention | Usual PC-MHI Care
Number analyzed (Participants) | 11 | 17
score on a scale
  GAD-7 total at Baseline | 12.5 (4.2) | 12.0 (3.1)
  GAD-7 total at Post (16 weeks) | 4.6 (5.2) | 9.1 (5.2)
Statistical Analysis 1: Comparison: Brief Anxiety Intervention vs Usual PC-MHI Care; comparisons of groups at post-assessment controls for baseline GAD-7 total scores; Test type: Superiority; p = 0.035, ANCOVA — a priori threshold for statistical significance was p<=.05

2. Secondary Outcome: Patient Health Questionnaire-9 at Post-Assessment
Description: The secondary outcome of depressive symptom severity will be measured by the Patient Health Questionnaire-9 (PHQ-9) self-report questionnaire, a validated measure that is widely used in VA primary care. Participants rate how often they have been bothered by each of 9 symptoms over the last 2 weeks on a Likert scale from 0 (not at all) to 3 (nearly every day). Scores are summed to create a total score from 0 to 27 indicating severity of depressive symptoms; higher scores indicate greater severity. The total score is sensitive to change from treatment. The PHQ-9 has demonstrated reliability and validity.
Time Frame: Baseline & Post-Assessment (at 16 weeks)
Population: Enrolled Participants who completed Post-Assessment at 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Anxiety Intervention | Usual PC-MHI Care
Number analyzed (Participants) | 11 | 17
score on a scale
  PHQ-9 total at Baseline | 10.5 (5.0) | 10.8 (5.2)
  PHQ-9 total at Post (16 weeks) | 5.1 (4.7) | 7.6 (6.4)
Statistical Analysis 1: Comparison: Brief Anxiety Intervention vs Usual PC-MHI Care; comparisons of groups at post-assessment controls for baseline PHQ-9 total scores; Test type: Superiority; p = 0.231, ANCOVA — a priori threshold for statistical significance was p<=0.05

3. Secondary Outcome: Depression Anxiety Stress Scale-21 Anxiety Subscale Change
Description: The secondary outcome of anxiety symptoms will be measured with the Depression Anxiety Stress Scale-21 (DASS-21) Anxiety Subscale. Participants indicate how much each of 7 items applies to them over the past week on a scale from 0 (did not apply to me at all) to 3 (applied to me very much, or most of the time). Scores are summed and multiplied by 2 to create a total score ranging from 0 to 42; higher scores indicate higher anxiety symptoms. This measure has good psychometric properties in both clinical and non-clinical samples. The DASS-21 reliably distinguishes between symptoms of anxiety (panic/worry), stress (tension/agitation), and depression (low mood/anhedonia), which are highly comorbid.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks, & Post-Assessment (at 16 weeks)
Population: Enrolled participants who completed each assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Anxiety Intervention | Usual PC-MHI Care
Number analyzed (Participants) | 17 | 18
score on a scale
  DASS-21 Anxiety subscale total at Baseline | 12.4 (9.4) | 10.1 (9.5)
  DASS-21 Anxiety subscale total at 4 weeks: number analyzed (Participants) | 16 | 18
  DASS-21 Anxiety subscale total at 4 weeks | 10.4 (7.3) | 9.4 (8.3)
  DASS-21 Anxiety subscale total at 8 weeks: number analyzed (Participants) | 14 | 18
  DASS-21 Anxiety subscale total at 8 weeks | 7.0 (6.3) | 10.1 (8.6)
  DASS-21 Anxiety subscale total at 12 weeks: number analyzed (Participants) | 13 | 17
  DASS-21 Anxiety subscale total at 12 weeks | 4.8 (4.7) | 9.9 (7.4)
  DASS-21 Anxiety subscale total at Post Assessment (16 weeks): number analyzed (Participants) | 11 | 17
  DASS-21 Anxiety subscale total at Post Assessment (16 weeks) | 4.9 (5.0) | 9.6 (7.7)
Statistical Analysis 1: Comparison: Brief Anxiety Intervention vs Usual PC-MHI Care; Change in DASS-21 Anxiety subscale total from Baseline to 4 weeks; Test type: Superiority — Testing null hypothesis of no difference between groups; p = 0.393, Mixed Models Analysis — a priori threshold for statistical significance was p<=0.05
Statistical Analysis 2: Comparison: Brief Anxiety Intervention vs Usual PC-MHI Care; Change in DASS-21 Anxiety subscale total from Baseline to 8 weeks; Test type: Superiority — Testing null hypothesis of no difference between groups; p = 0.022, Mixed Models Analysis — a priori threshold for statistical significance was p<=0.05
Statistical Analysis 3: Comparison: Brief Anxiety Intervention vs Usual PC-MHI Care; Change in DASS-21 Anxiety subscale total from Baseline to 12 weeks; Test type: Superiority — Testing null hypothesis of no difference between groups; p = 0.013, Mixed Models Analysis — a priori threshold for statistical significance was p<=0.05
Statistical Analysis 4: Comparison: Brief Anxiety Intervention vs Usual PC-MHI Care; Change in DASS-21 Anxiety subscale total from Baseline to Post assessment (16 weeks); Test type: Superiority — Testing null hypothesis of no difference between groups; p = 0.049, Mixed Models Analysis — a priori threshold for statistical significance was p<=0.05

4. Secondary Outcome: Depression Anxiety Stress Scale-21 Depression Subscale Change
Description: The secondary outcome of depression symptoms will be measured with the Depression Anxiety Stress Scale-21 (DASS-21) Depression Subscale. Participants indicate how much each of 7 items applies to them over the past week on a scale from 0 (did not apply to me at all) to 3 (applied to me very much, or most of the time). Scores are summed and multiplied by 2 to create a total score ranging from 0 to 42; higher scores indicate higher depressive symptoms. This measure has good psychometric properties in both clinical and non-clinical samples. The DASS-21 reliably distinguishes between symptoms of anxiety (panic/worry), stress (tension/agitation), and depression (low mood/anhedonia) which are highly comorbid.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks, & Post-Assessment (at 16 weeks)
Population: Enrolled participants who completed each assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Anxiety Intervention | Usual PC-MHI Care
Number analyzed (Participants) | 17 | 18
score on a scale
  DASS-21 Depression subscale total at Baseline | 15.6 (9.9) | 12.2 (9.5)
  DASS-21 Depression subscale total at 4 weeks: number analyzed (Participants) | 16 | 18
  DASS-21 Depression subscale total at 4 weeks | 8.1 (5.6) | 11.1 (11.2)
  DASS-21 Depression subscale total at 8 weeks: number analyzed (Participants) | 14 | 18
  DASS-21 Depression subscale total at 8 weeks | 6.0 (4.8) | 11.9 (9.6)
  DASS-21 Depression subscale total at 12 weeks: number analyzed (Participants) | 13 | 17
  DASS-21 Depression subscale total at 12 weeks | 4.5 (4.3) | 10.8 (10.8)
  DASS-21 Depression subscale total at Post-assessment (16 weeks): number analyzed (Participants) | 11 | 17
  DASS-21 Depression subscale total at Post-assessment (16 weeks) | 4.9 (4.9) | 9.9 (12.6)
Statistical Analysis 1: Comparison: Brief Anxiety Intervention vs Usual PC-MHI Care; Change in DASS-21 Depression subscale total from Baseline to 4 weeks; Test type: Superiority — Testing null hypothesis of no difference between groups; p = 0.008, Mixed Models Analysis — a priori threshold for statistical significance was p<=0.05
Statistical Analysis 2: Comparison: Brief Anxiety Intervention vs Usual PC-MHI Care; Change in DASS-21 Depression subscale total from Baseline to 8 weeks; Test type: Superiority — Testing null hypothesis of no difference between groups; p < 0.001, Mixed Models Analysis — a priori threshold for statistical significance was p<=0.05
Statistical Analysis 3: Comparison: Brief Anxiety Intervention vs Usual PC-MHI Care; Change in DASS-21 Depression subscale total from Baseline to 12 weeks; Test type: Superiority — Testing null hypothesis of no difference between groups; p < 0.001, Mixed Models Analysis — a priori threshold for statistical significance was p<=0.05
Statistical Analysis 4: Comparison: Brief Anxiety Intervention vs Usual PC-MHI Care; Change in DASS-21 Depression subscale total from Baseline to Post-assessment (16 weeks); Test type: Superiority — Testing null hypothesis of no difference between groups; p = 0.008, Mixed Models Analysis — a priori threshold for statistical significance was p<=0.05

5. Secondary Outcome: Depression Anxiety Stress Scale-21 Stress Subscale Change
Description: The secondary outcome of stress symptoms will be measured with the Depression Anxiety Stress Scale-21 (DASS-21) Stress Subscale. Participants indicate how much each of 7 items applies to them over the past week on a scale from 0 (did not apply to me at all) to 3 (applied to me very much, or most of the time). Scores are summed and multiplied by 2 to create a total score ranging from 0 to 42; higher scores indicate higher stress symptoms. This measure has good psychometric properties in both clinical and non-clinical samples. The DASS-21 reliably distinguishes between symptoms of anxiety (panic/worry), stress (tension/agitation), and depression (low mood/anhedonia), which are highly comorbid.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks, & Post-Assessment (at 16 weeks)
Population: Enrolled participants who completed each assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Anxiety Intervention | Usual PC-MHI Care
Number analyzed (Participants) | 17 | 18
score on a scale
  DASS-21 Stress subscale total at Baseline | 18.7 (8.6) | 17.8 (6.9)
  DASS-21 Stress subscale total at 4 weeks: number analyzed (Participants) | 16 | 18
  DASS-21 Stress subscale total at 4 weeks | 16.9 (8.0) | 17.3 (11.2)
  DASS-21 Stress subscale total at 8 weeks: number analyzed (Participants) | 14 | 18
  DASS-21 Stress subscale total at 8 weeks | 11.7 (6.9) | 17.0 (10.4)
  DASS-21 Stress subscale total at 12 weeks: number analyzed (Participants) | 13 | 17
  DASS-21 Stress subscale total at 12 weeks | 10.5 (8.0) | 16.4 (11.0)
  DASS-21 Stress subscale total at Post-assessment (16 weeks): number analyzed (Participants) | 11 | 17
  DASS-21 Stress subscale total at Post-assessment (16 weeks) | 7.6 (9.2) | 14.1 (10.3)
Statistical Analysis 1: Comparison: Brief Anxiety Intervention vs Usual PC-MHI Care; Change in DASS-21 Stress subscale total from Baseline to 4 weeks; Test type: Superiority — Testing null hypothesis of no difference between groups; p = 0.440, Mixed Models Analysis — a priori threshold for statistical significance was p<=0.05
Statistical Analysis 2: Comparison: Brief Anxiety Intervention vs Usual PC-MHI Care; Change in DASS-21 Stress subscale total from Baseline to 8 weeks; Test type: Superiority — Testing null hypothesis of no difference between groups; p = 0.022, Mixed Models Analysis — a priori threshold for statistical significance was p<=0.05
Statistical Analysis 3: Comparison: Brief Anxiety Intervention vs Usual PC-MHI Care; Change in DASS-21 Stress subscale total from Baseline to 12 weeks; Test type: Superiority — Testing null hypothesis of no difference between groups; p = 0.032, Mixed Models Analysis — a priori threshold for statistical significance was p<=0.05
Statistical Analysis 4: Comparison: Brief Anxiety Intervention vs Usual PC-MHI Care; Change in DASS-21 Stress subscale total from Baseline to Post-assessment (16 weeks); Test type: Superiority — Testing null hypothesis of no difference between groups; p = 0.091, Mixed Models Analysis — a priori threshold for statistical significance was p<=0.05

6. Secondary Outcome: Overall Anxiety Severity and Impairment Scale Change
Description: Functional impairment from anxiety symptoms will be measured using the Overall Anxiety Severity and Impairment Scale (OASIS), which measures symptom severity and functional impairment across anxiety disorders and subthreshold symptoms. The 5-item scale demonstrates reliability (Cronbach's alpha = .84 in primary care sample) and validity in primary care patients. Participants indicate the frequency and intensity of anxiety, level of avoidance, and interference with activities and social functioning on a Likert scale from 0 to 4. Scores are summed to create a total score ranging from 0 to 20; higher scores indicate greater symptom severity and functional impairment from anxiety.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks, & Post-Assessment (at 16 weeks)
Population: Enrolled participants who completed each assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Anxiety Intervention | Usual PC-MHI Care
Number analyzed (Participants) | 17 | 18
score on a scale
  OASIS total at Baseline | 9.4 (3.9) | 9.4 (2.8)
  OASIS total at 4 weeks: number analyzed (Participants) | 16 | 18
  OASIS total at 4 weeks | 6.2 (3.3) | 8.2 (3.8)
  OASIS total at 8 weeks: number analyzed (Participants) | 14 | 18
  OASIS total at 8 weeks | 5.5 (3.4) | 8.0 (4.6)
  OASIS total at 12 weeks: number analyzed (Participants) | 13 | 17
  OASIS total at 12 weeks | 4.8 (3.7) | 8.2 (4.0)
  OASIS total at Post-assessment (16 weeks): number analyzed (Participants) | 11 | 17
  OASIS total at Post-assessment (16 weeks) | 4.1 (3.8) | 7.4 (3.8)
Statistical Analysis 1: Comparison: Brief Anxiety Intervention vs Usual PC-MHI Care; Change in OASIS total score from Baseline to 4 weeks; Test type: Superiority — Testing null hypothesis of no difference between groups; p = 0.058, Mixed Models Analysis — a priori threshold for statistical significance was p<=0.05
Statistical Analysis 2: Comparison: Brief Anxiety Intervention vs Usual PC-MHI Care; Change in OASIS total score from Baseline to 8 weeks; Test type: Superiority — Testing null hypothesis of no difference between groups; p = 0.032, Mixed Models Analysis — a priori threshold for statistical significance was p<=0.05
Statistical Analysis 3: Comparison: Brief Anxiety Intervention vs Usual PC-MHI Care; Change in OASIS total score from Baseline to 12 weeks; Test type: Superiority — Testing null hypothesis of no difference between groups; p = 0.007, Mixed Models Analysis — a priori threshold for statistical significance was p<=0.05
Statistical Analysis 4: Comparison: Brief Anxiety Intervention vs Usual PC-MHI Care; Change in OASIS total score from Baseline to Post assessment (16 weeks); Test type: Superiority — Testing null hypothesis of no difference between groups; p = 0.044, Mixed Models Analysis — a priori threshold for statistical significance was p<=0.05

7. Secondary Outcome: Overall Depression Severity and Impairment Scale Change
Description: Functional impairment from depressive symptoms will be measured using the Overall Depression Severity and Impairment Scale (ODSIS), which measures symptom severity and functional impairment across depressive disorders and subthreshold symptoms. Adapted from the OASIS to apply to depression, the 5-item scale demonstrates reliability (Cronbach's alpha = .92 in community sample of adults) and validity. Participants indicate the frequency and intensity of depressive symptoms, difficulty engaging in activities, and interference with work/school/home activities and social functioning on a Likert scale from 0 to 4. Scores are summed to create a total score ranging from 0 to 20; higher scores indicate greater symptom severity and functional impairment due to depression.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks, & Post-Assessment (at 16 weeks)
Population: Enrolled participants who completed each assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Anxiety Intervention | Usual PC-MHI Care
Number analyzed (Participants) | 17 | 18
score on a scale
  ODSIS total at Baseline | 6.5 (4.3) | 6.2 (4.5)
  ODSIS total at 4 weeks: number analyzed (Participants) | 16 | 18
  ODSIS total at 4 weeks | 4.3 (3.7) | 5.3 (4.4)
  ODSIS total at 8 weeks: number analyzed (Participants) | 14 | 18
  ODSIS total at 8 weeks | 3.9 (3.5) | 5.6 (5.5)
  ODSIS total at 12 weeks: number analyzed (Participants) | 13 | 17
  ODSIS total at 12 weeks | 2.7 (3.3) | 6.2 (5.3)
  ODSIS total at Post-assessment (16 weeks): number analyzed (Participants) | 11 | 17
  ODSIS total at Post-assessment (16 weeks) | 3.0 (3.7) | 5.0 (4.8)
Statistical Analysis 1: Comparison: Brief Anxiety Intervention vs Usual PC-MHI Care; Change in ODSIS total from Baseline to 4 weeks; Test type: Superiority — Testing null hypothesis of no difference between groups; p = 0.328, Mixed Models Analysis — a priori threshold for statistical significance was p<=0.05
Statistical Analysis 2: Comparison: Brief Anxiety Intervention vs Usual PC-MHI Care; Change in ODSIS total from Baseline to 8 weeks; Test type: Superiority — Testing null hypothesis of no difference between groups; p = 0.148, Mixed Models Analysis — a priori threshold for statistical significance was p<=0.05
Statistical Analysis 3: Comparison: Brief Anxiety Intervention vs Usual PC-MHI Care; Change in ODSIS total from Baseline to 12 weeks; Test type: Superiority — Testing null hypothesis of no difference between groups; p = 0.002, Mixed Models Analysis — a priori threshold for statistical significance was p<=0.05
Statistical Analysis 4: Comparison: Brief Anxiety Intervention vs Usual PC-MHI Care; Change in ODSIS total from Baseline to Post-assessment (16 weeks); Test type: Superiority — Testing null hypothesis of no difference between groups; p = 0.069, Mixed Models Analysis — a priori threshold for statistical significance was p<=0.05

8. Other Pre Specified Outcome: Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form at Post-Assessment
Description: Quality of life will be measured using the Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q-LES-Q-SF), which measures overall enjoyment and satisfaction with various aspects of life. The 16-item scale is reliable (alpha = .86) and valid. Participants rate satisfaction with each domain on a Likert scale from 1 to 5. Scores for items 1-14 are summed to create a total score ranging from 14 to 70; higher scores indicate higher quality of life.
Time Frame: Baseline & Post-Assessment (at 16 weeks)
Population: Enrolled Participants who completed Post-Assessment at 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Anxiety Intervention | Usual PC-MHI Care
Number analyzed (Participants) | 11 | 17
score on a scale
  Q-LES-Q-SF total at Baseline | 44.9 (8.5) | 43.8 (7.4)
  Q-LES-Q-SF total at Post (16 weeks) | 49.9 (8.1) | 48.7 (10.0)
Statistical Analysis 1: Comparison: Brief Anxiety Intervention vs Usual PC-MHI Care; comparisons of groups at post-assessment controls for baseline Q-LES-Q-SF total scores; Test type: Superiority; p = 0.928, ANCOVA — a priori threshold for statistical significance was p<=0.05

9. Other Pre Specified Outcome: Engagement in Treatment
Description: This feasibility outcome measure is the number who attended one or more treatment sessions
Time Frame: Post-assessment (16 weeks)
Population: All participants who enrolled in the study
Measure: Number; unit: participants
Arm/Group | Brief Anxiety Intervention | Usual PC-MHI Care
Number analyzed (Participants) | 17 | 18
participants | 15 | 13
Statistical Analysis 1: Comparison: Brief Anxiety Intervention vs Usual PC-MHI Care; Testing null hypothesis of no difference between groups; Test type: Superiority; p = 0.402, Fisher Exact — a priori threshold for statistical significance was p<.05; degrees of freedom = 1

10. Other Pre Specified Outcome: Number of Treatment Sessions Completed
Description: This feasibility measure is the number of treatment sessions completed during the 16-week active treatment phase
Time Frame: Post-assessment (16 weeks)
Population: All participants enrolled in the study
Measure: Mean (Standard Deviation); unit: sessions
Arm/Group | Brief Anxiety Intervention | Usual PC-MHI Care
Number analyzed (Participants) | 17 | 18
sessions | 4.7 (2.2) | 1.8 (1.6)
Statistical Analysis 1: Comparison: Brief Anxiety Intervention vs Usual PC-MHI Care; Testing the null hypothesis of no difference between groups; Test type: Superiority; p < 0.001, t-test, 2 sided — a priori threshold for statistical significance was p<=.05

11. Other Pre Specified Outcome: Treatment Satisfaction
Description: The acceptability outcome of treatment satisfaction was assessed using the 8-item version of the Client Satisfaction Questionnaire. This self-report questionnaire has evidence of reliability and validity. Participants indicate their agreement with 8 items on a 4-point Likert scale. Scores are summed to create a total score ranging from 8 to 32; higher scores indicate greater satisfaction with treatment.
Time Frame: Post-assessment (at 16 weeks)
Population: All participants who completed the Post-assessment (at 16 weeks) and reported attending at least one treatment session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Anxiety Intervention | Usual PC-MHI Care
Number analyzed (Participants) | 10 | 13
score on a scale | 29.80 (2.82) | 24.23 (5.69)
Statistical Analysis 1: Comparison: Brief Anxiety Intervention vs Usual PC-MHI Care; Testing the null hypothesis of no difference between groups; Test type: Superiority; p = .006, t-test, 2 sided — a priori threshold for statistical significance was p<=.05; Used Satterthwaite method given unequal variances

12. Other Pre Specified Outcome: Treatment Credibility
Description: The acceptability outcome of treatment credibility was measured using a 4-item adapted version of the Expectancy Rating Scale, which asks patients to rate, on a Likert scale from 0 (not at all) to 10 (extremely), how logical this type of anxiety treatment seems, how confident they are that the treatment would eliminate anxiety, how confident they would be in recommending the treatment to a friend with anxiety, and how much improvement they expect to result from it. Scores are summed to create a total score ranging from 0 to 40; higher scores indicate greater treatment credibility.
Time Frame: Post-assessment (16 weeks)
Population: All participants who completed the Post-assessment (at 16 weeks) and reported attending at least one treatment session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Anxiety Intervention | Usual PC-MHI Care
Number analyzed (Participants) | 10 | 13
score on a scale | 34.20 (5.51) | 22.31 (11.49)
Statistical Analysis 1: Comparison: Brief Anxiety Intervention vs Usual PC-MHI Care; Testing the null hypothesis of no difference between groups; Test type: Superiority; p = 0.004, t-test, 2 sided — a priori threshold for statistical significance was p<=.05; used Satterthwaite method given unequal variances

13. Other Pre Specified Outcome: Therapeutic Alliance
Description: The acceptability outcome of therapeutic alliance was measured using the 12-item Working Alliance Inventory-Short Form Revised, which asks patients to rate, on a Likert scale from 1 (seldom) to 5 (always), their experience of the therapist in terms of quality of the relationship bond, agreement on the goals of treatment, and agreement on the tasks of treatment. Scores are summed to create a total score ranging from 12 to 60. This measure has good reliability and validity.
Time Frame: Post-assessment (16 weeks)
Population: All participants who completed Post-assessment (16 weeks) and reported attending at least one treatment session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Anxiety Intervention | Usual PC-MHI Care
Number analyzed (Participants) | 10 | 13
score on a scale | 55.00 (5.54) | 42.62 (9.73)
Statistical Analysis 1: Comparison: Brief Anxiety Intervention vs Usual PC-MHI Care; Testing the null hypothesis of no difference between groups; Test type: Superiority; p = 0.002, t-test, 2 sided — a priori threshold for statistical significance was p<=.05

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the course of a participant's study participation, 16 weeks.
Description: n/a (same definitions as clinicaltrials.gov). Adverse event collection included systematic assessment (e.g., anxiety and depressive symptoms assessed at each treatment session in intervention condition and at each study assessment) and non-systematic assessment (e.g., participant self-report, information in participant medical record).
Arm/Group | Brief Anxiety Intervention | Usual PC-MHI Care
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/17 | 1/18
Other Adverse Events (participants affected / at risk) | 1/17 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brief Anxiety Intervention (N=17) | Usual PC-MHI Care (N=18)
Hospitalization (Cardiac disorders) | 0 (0) | 1 (1) — Participant was admitted to the hospital overnight for monitoring of a pre-existing medical condition that was unrelated to the treatment received in the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brief Anxiety Intervention (N=17) | Usual PC-MHI Care (N=18)
Symptom exacerbation (Social circumstances) | 1 (1) | 0 (0) — Clinically significant increase in anxiety and depression symptom severity from 2nd to 3rd intervention session. This was unrelated to the intervention or study, rather it was directly related to a psychosocial stressor (father unexpectedly died).

LIMITATIONS AND CAVEATS:
This was a single-site pilot trial with a small sample size so results should be interpreted with caution. The attrition rate for assessments was slightly higher in the intervention (vs. comparison) condition. However, multi-level modeling analyses made use of all participant data provided. We did not have a follow-up assessment to examine whether treatment gains were maintained over time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/89/NCT03794089/Prot_SAP_000.pdf